CLINICAL TRIAL: NCT03715127
Title: Phase II, Randomized, Double Blind, Placebo Controlled, Parallel Group, Single Center Study of Psilocybin Efficacy in Major Depression
Brief Title: Clinical, Neurocognitive, and Emotional Effects of Psilocybin in Depressed Patients - Proof of Concept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Schweizerischer Nationalfonds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSIDEPR128
Record Dates: First submitted 2018-10-16; First posted 2018-10-22 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; 5HT-2A; Psilocybin; clinical efficacy; self; emotion regulation; placebo-controlled; proof-of-concept
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Emotional Regulation | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: placebo-controlled, quadruple-blind, randomized, mono-centric
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: quadruple-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): one oral dose of 100% mannitol (placebo)
  Interventions: Drug: Placebo oral capsule
- Psilocybin (Active Comparator): one oral dose of 0.215mg/kg psilocybin (verum)
  Interventions: Drug: Psilocybine oral capsule

INTERVENTIONS:
Drug: Psilocybine oral capsule — single dose of psilocybin (0.215mg / kg body weight)
  Arms: Psilocybin
Drug: Placebo oral capsule — single dose of placebo (100% mannitol)
  Arms: Placebo

SUMMARY:
Effects of serotonin 2A/1A receptor stimulation by psilocybin on mood and emotion processing in major depressive disorder: a randomized double-blind placebo-controlled study

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is one of the world's greatest contributor to the global burden of disease and MDD affects around 17% of the Swiss population (Tomonaga et al. 2013). It is a chronic condition and can cause the affected person to suffer greatly and function poorly at work, at school and in the family. More than 1'000 suicides were recorded in Switzerland in 2014, about 90% of these fatalities were related to depression or other psychiatric problems. Suicide is the second leading cause of death in individuals 15-24 years of age (Insel & Charney 2003).

Current pharmacotherapies, including monoaminergic-acting antidepressants, require prolonged administration (weeks if not months) for clinical improvement. This lag time, as well as a high non-response rate, emphasizes the need for better and faster-acting antidepressant medications. However, psychopharmacological research has largely failed to produce novel and more efficacious treatment options for MDD since decades. Advanced pharmaceutical antidepressants should ideally facilitate the psychotherapeutic process for patients, reduce the time onset of antidepressant efficacy, and prime neuroplastic adaptations relevant to symptom improvement. Such novel therapeutics are much needed and would address this detrimental public health problem, particularly in treatment-resistant patients.

Early clinical studies using the psychotropic compound psilocybin (4-phosphoryloxy-N,N-dimethyltryptamine) as an adjunct in psychotherapy reported a significant improvement of clinical symptoms in depression and anxiety disorder (Leuner 1961, 1981). Psilocybin is the main psychoactive principle of the group of hallucinogenic fungi (Hofmann 1968), commonly known as magic mushrooms, and acts as partial agonist at cortical and sub-cortical serotonin 5-HT2A and 5-HT1A receptors. At moderate doses, psilocybin produces a dream-like state of consciousness (Kraehenmann et al. 2016) characterized by perceptual alterations, enhanced mood, facilitated autobiographic memory recollection, and a change of perspective on the self (Leuner 1981; Studerus et al. 2011). Recent clinical studies applying placebo-controlled designs support and extend these early findings by showing that a single dose of psilocybin leads to a fast and sustained reduction in anxiety and depression as well as an improvement of quality of life in advanced cancer patients (Griffiths 2015, Grob et al. 2011). Furthermore, a recent open-label feasibility study showed rapid-onset, sustained symptom improvements over 3 weeks in a small sample of treatment-resistant depressed patients following two psilocybin treatment sessions (Carhart-Harris et al. 2016). Accumulating evidence from pharmacological and neuroimaging studies suggests that psilocybin may produce its antidepressant effects via activation of 5-HT2A receptors located in prefrontal-limbic structures that are also implicated in the pathophysiology of depression (Kraehenmann & Vollenweider et al. 2015; Vollenweider und Kometer 2010; Disner et al. 2011). In addition, molecular studies suggest that the enduring symptom improvement after a single dose of psilocybin may be mediated through downstream effects on the glutamate system and a subsequent activation of neuroplastic factors such as brain-derived neurotrophic factor (BDNF) (Catlow et al. 2013, Barre et al. 2016).

The present clinical trial aims at investigating the putative antidepressant effects of a single moderate dose of psilocybin (0.215 mg/kg) in patients suffering from MDD by applying a randomized, double-blind, placebo-controlled design. The specific aims of this project are: 1. To investigate whether psilocybin in combination with short-term focused psychotherapy will reduce core symptoms in patients with MDD. 2. Using functional magnetic resonance imaging (fMRI) to longitudinally assess whether a single dose of psilocybin will post-acutely change the negative emotion processing bias in patients with MDD and whether the change in emotion processing bias will predict subsequent symptom improvement. In addition, the investigators will analyze whether psilocybin will lead to sustained changes in functional neuronal network connectivity (FC), e.g. in amygdala-prefrontal FC. 3. To investigate whether psilocybin will increase BDNF plasma concentration and whether the change in BDNF is related to changes in fMRI markers and the subsequent mood improvement.

Recent reviews indicate that impaired neuroplasticity is at the core of the pathophysiology moods and stress-related disorders. Current available antidepressants have been developed with the aim of providing symptom relief rather than targeting neuroplastic impairments. In contrast to this, the present proposal builds on promising new findings that single dose of psilocybin, presumably via a 5-HT2A receptor driven glutamatergic mechanism, leads to a rapid enhancement in neuronal resilience and a to a change in the function of neuronal networks underlying depressive symptoms and behavior. Targeting neuroplasticity with such novel approaches appears to be important for reversing cognitive schemata and emotion processing biases, fostering enduring improvements in mood and cognitive flexibility (Krystal et al. 2009).

Expected value: this is the first randomized, double-blind, placebo-controlled clinical trial (RCT) of psilocybin treatment in MDD. Using state-of-the art behavioral, neuroimaging, and neuroplasticity methodology, the results of this study will help elucidate urgently needed new treatment mechanisms in MDD. Should it turn out that a single moderate dose of psilocybin vs. placebo in conjunction with psychotherapy may rapidly and sustainedly reduce depressive symptoms, this will be a major breakthrough in finding a novel and fast acting treatment strategy in depressed patients. Therefore, the results of this study will have high impact on the field of pharmacological research into novel antidepressant medication.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Informed consent as documented by signature
* Male and female in- and outpatients 18 years to 60 years of age
* Right-handedness
* DSM-IV-diagnosis of mild or moderate major depressive episode without psychotic features (based on clinical assessment and confirmed by the SCID Interview)
* Score of ≥ 10 and ≤40 on the Montgomery-Asberg Depression Rating Scale (MADRS) at both screening and baseline visits.
* Drug free from any psychotropic medication for at least two weeks (or five weeks for fluoxetine) before enrolling in the study
* Judged clinically not to be a serious suicide risk
* Good physical health with no unstable medical conditions, as determined by medical history, physical examination, routine blood labs, electrocardiogram, urineanalysis, and urine toxicology
* Normal level of language comprehension and German or Swiss-German as first language
* Willing to refrain from drinking alcohol the day before testing days, from drinking alcohol and caffeinated drinks during the testing days and from consuming psychoactive substances 2 weeks before enrolling in the study and for the remainder of the study
* Women of childbearing potential must be using an effective, established method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices. Note: female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Have a family member or friend who can pick them up and stay with them overnight after the psilocybin administration sessions (driving is forbidden at drug treatment days)

Exclusion Criteria:

* Lifetime history of bipolar disorder (I, II, not otherwise specified)
* Lifetime history of schizophrenia, schizoaffective disorder, or psychosis not otherwise specified
* History of DSM-IV drug or alcohol dependence or abuse (except for caffeine or nicotine) within three months prior to enrollment
* Comorbid Axis I anxiety disorder diagnoses will be permitted if they do not require current treatment
* Family history of schizophrenia or schizoaffective disorder, or bipolar disorder type 1 (first or second degree relatives)
* Lifetime history of hallucinogen use on more than 10 occasions
* Getting psychotherapeutic or psychological treatment from third parties during the study is forbidden
* Abnormal electrocardiogram
* Any unstable illness as determined by history or laboratory tests
* BMI <17 or >35
* Uncorrected hypo- or hyperthyroidism
* Women who are pregnant or breast feeding, or have the intention to become pregnant during the course of the study
* Contraindications to magnetic resonance imaging (MRI safety form)
* During the study, new use or dose changes of already existing concomitant medication without prior informing the investigators is forbidden
* Allergy, hypersensitivity, or other adverse reaction to previous use of psilocybin or other hallucinogens
* High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support)
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Scale | Day 32
  observer-rated score for depression
Beck Depression Inventory | Day 32
  self-rated score for depression

SECONDARY OUTCOMES:
Changes in BOLD signal over time as measured by fMRI | Day 17, 20, 32
  3 times assessement of fMRI
5 Dimensions- Altered States of consciousness(5D-ASC) | Day 18
  Assessment of subjective alterations in state of conciousness

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jungwirth J, von Rotz R, Dziobek I, Vollenweider FX, Preller KH. Psilocybin increases emotional empathy in patients with major depression. Mol Psychiatry. 2025 Jun;30(6):2665-2672. doi: 10.1038/s41380-024-02875-0. Epub 2024 Dec 18. PMID 39695323
- [Derived] von Rotz R, Schindowski EM, Jungwirth J, Schuldt A, Rieser NM, Zahoranszky K, Seifritz E, Nowak A, Nowak P, Jancke L, Preller KH, Vollenweider FX. Single-dose psilocybin-assisted therapy in major depressive disorder: A placebo-controlled, double-blind, randomised clinical trial. EClinicalMedicine. 2022 Dec 28;56:101809. doi: 10.1016/j.eclinm.2022.101809. eCollection 2023 Feb. PMID 36636296